CLINICAL TRIAL: NCT05248802
Title: Randomized Controlled Trial of DLBS2411 Treatment For Functional Dyspepsia
Brief Title: DLBS2411 Treatment For Functional Dyspepsia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS2411-0419
Record Dates: First submitted 2022-01-26; First posted 2022-02-21 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; DLBS2411; Epigastric Pain Syndrome; Postprandial Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Placebo DLBS2411 2 x 1 caplet daily, given everyday for 4 weeks of study period
  Interventions: Drug: Placebo caplet of DLBS2411
- DLBS2411 (Experimental): DLBS2411 caplet 2 x 250 mg daily, given everyday for 4 weeks of study period
  Interventions: Drug: DLBS2411

INTERVENTIONS:
Drug: Placebo caplet of DLBS2411 — 1 caplet of placebo DLBS2411, twice daily
  Other Names: Placebo caplet of Redacid
  Arms: Control
Drug: DLBS2411 — 1 caplet of DLBS2411 250 mg, twice daily
  Other Names: Redacid
  Arms: DLBS2411

SUMMARY:
This is a 2-arm, prospective, double-blind, randomized and placebo-controlled study using DLBS2411 at a dose of 250 mg twice daily (before morning and evening meals), for a 4-week course of therapy, for the treatment of patients with functional dyspepsia (FD), and an additional 8 weeks after end of therapy (Week 12) for follow-up visit.

The bioactive fraction of DLBS2411 has been proved at cellular and genetic levels to have an antiulcer effect through both suppressing the gastric acidity and enhancing gastric mucosal protection. The anti-secretory effect of DLBS2411 is exerted through the inhibition of H+/K+ ATPase 'pump' as well as down-regulation of the H+/K+ ATPase gene expression, thus suppressing gastric acid secretion; while its cytoprotective defense mechanism works through the promotion of cyclooxygenase-2 (COX-2) derived prostaglandin (PgE2) synthesis, thus promoting gastrointestinal submucosal blood-flow, stimulating secretion of gastric-epithelial mucous and bicarbonate; anti-oxidative activity; and endothelial-nitric oxide (NO) formation. The mechanism altogether demonstrated DLBS2411's protective capacity to the gastric and colon mucosa by promoting mucous synthesis and stimulating mucosal blood flow.

Having such mechanisms of action, DLBS2411 is hypothesized to benefit subjects with gastric acid disorders such as in functional dyspepsia, gastro-intestinal reflux disease (GERD), peptic-ulcer, and irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
Study population will be patients with functional dyspepsia (FD) who come to the study site. There will be 100 subjects (50 subjects in each group) planned to be enrolled in the study.

There will be 2 groups of treatment; Treatment 1: placebo DLBS2411 caplet Treatment 2: DLBS2411 250 mg caplet Each study medication will be administered 1 caplet twice daily, 30 minutes before meal, in the morning and evening.

Eligible subjects will be randomly allocated to receive either Treatment 1 or Treatment 2 for 4 weeks, in a double blind fashion. Subjects will be instructed to come to the clinic every 2-week interval throughout the 4-week study period (at Week 2, and 4, respectively) and 8 weeks after the end of therapy (Week 12), for efficacy evaluation. The safety evaluation will be performed at Baseline and End of therapy (Week 4). Adverse events will be monitored at baseline and every follow-up visit including End of study (Week 12).

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent prior to participation in the study.
2. Male or female subjects aged of 18 - 75 years old.
3. Meet Rome IV criteria for FD, which includes:

   1. One or more of the following symptoms:

      * bothersome postprandial fullness
      * early satiation, that prevents finishing a regular meal, at least several times per week.
      * epigastric pain, epigastric burning. The symptoms are persistently present (i.e. occurring at least one day per month (for male) or 2-3 days per month (for female) for at least the past 3 months with symptom onset at least 6 months prior to study Screening.
   2. Having no evidence of structural or organic gastrointestinal (GI) disease that is likely to explain the symptoms, as verified by a normal esophagogastroduodenoscopy (EGD) performed within the past 3 years.
4. Subjects who tested negative for Helicobacter pylori by urea breath-test, histological or rapid test during the screening period.
5. Able to take oral medication.

Key Exclusion Criteria:

1. Pregnancy, breast-feeding females.
2. Subjects suspected COVID-19 by clinical symptoms and rapid antigen test (reactive result) for SARS-COV-2.
3. GERD as confirmed by any documented history of endoscopic esophagitis, or clinical symptoms such as predominant heartburn or acid regurgitation, >2x/week in the prior year.
4. History of or known or suspected Zollinger Ellison syndrome.
5. History of or known gastrointestinal malignancy or ulcers associated to malignancy.
6. Hepatic cirrhosis or abnormal liver laboratory findings (defined as >3xULN of ALT or AST).
7. Being under hemodialysis therapy or having advanced chronic kidney disease (defined as eGFR <60 mL/min).
8. History of or known congestive heart failure NYHA class III and IV, or any other uncontrolled chronic diseases, such as: uncontrolled hypertension (systolic/diastolic blood pressure ≥160/100 mmHg); uncontrolled diabetes (HbA1c c ≥7%).
9. Currently known being afflicted by serious infection(s), or any known severe illness(es) which are judged by the Investigator could interfere with subjects' safety and/or study evaluation.
10. Taking medication affecting the gastrointestinal system within 2 weeks prior to Screening, such as: prokinetics, acid release inhibitors (histamine-2-receptor [H2]- antagonists, proton pump inhibitors [PPI], or potassium-competitive acid blockers), gastric mucosa protectors (sucralfate, rebamipide), and any gastric-relevant herbal medicines.
11. Participation in any other clinical studies within 30 days prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Short-Form Nepean Dyspepsia Index (SF-NDI) | Week 4
  Change of disease specific quality of life as measured by short-form NDI (SF-NDI) after 4 weeks of therapy (Week 4).
  The SF-NDI consists of 10 quality-of-life (QoL)-items, each of which is measured by 5-point Likert scales from 0 (not at all or not applicable), 1 (a little), 2 (moderately), 3 (quite a lot) to 4 (extremely). The lower score indicates an improved outcome.

SECONDARY OUTCOMES:
Short-Form Nepean Dyspepsia Index (SF-NDI) | Week 2 and 12
  Change of disease specific quality of life as measured by short-form NDI (SF-NDI) after 2 weeks of therapy (Week 2) and additional 8 weeks after end of therapy (Week 12).
  The SF-NDI consists of 10 quality-of-life (QoL)-items, each of which is measured by 5-point Likert scales from 0 (not at all or not applicable), 1 (a little), 2 (moderately), 3 (quite a lot) to 4 (extremely). The lower score indicates an improved outcome.
Visual Analogue Scale (VAS) | Week 2, 4, and 12
  Change of the individual symptom intensity as indicated by Visual Analogue Scale (VAS) reduction after 2 and 4 weeks of therapy and 8 weeks after the end of therapy (Week 2, 4 and 12, respectively).
  The VAS of pain intensity is rated from 0 to 100 on a 100-mm line, with the end points indicating: no pain (0) and the worst pain it could possible be (100).
The proportion of subjects reaching adequate / satisfactory relief from FD symptoms | Week 2, 4, and 12
  The proportion of subjects reaching adequate / satisfactory relief from FD symptoms based on subjects" subjective evaluation on overall symptom relief at Week 2, Week 4 and additional 8 weeks after end of therapy (Week 12)
Number of adverse event during the study | Week 2, 4, and 12
  Number of adverse event during the study will be observed throughout the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Ari F Syam, Prof, MD, Sp.PD-KGEH, Principal Investigator — Division of Gastroenterology Department of Internal Medicine Faculty of Medicine, University of Indonesia Dr. Cipto Mangunkusumo National General Hospital, Jakarta Indonesia; Agasjtya W Wardhana, MD, Sp.PD-KGEH, Principal Investigator — Department of Internal Medicine Budhi Asih Hospital, East Jakarta, Indonesia; Nugroho B Santoso, MD, Sp.PD, Principal Investigator — Department of Internal Medicine Pasar Rebo Hospital, South Jakarta, Indonesia; Hery D Purnomo, Dr, MD, Sp.PD-KGEH, Principal Investigator — Department of Internal Medicine Dr. Kariadi General Hospital, Semarang, Indonesia; Triyanta Y Pramana, Dr, MD, Sp.PD-KGEH, Principal Investigator — Department of Internal Medicine Dr. Moewardi Hospital, Surakarta, Indonesia; Mulyana Edi, MD, Sp.PD-KGEH, Principal Investigator — Department of Internal Medicine Fatmawati General Hospital, Jakarta,; Coana Sukmagautama, MD, Sp.PD, M.Kes., Principal Investigator — Department of Internal Medicine Universitas Sebelas Maret (UNS) Hospital, Sukoharjo, Indonesia; Ulfa Kholili, MD, Sp.PD-KGEH, Principal Investigator — Department of Internal Medicine, Dr. Soetomo General Hospital, Surabaya, Indonesia
Locations (8):
- Indonesia (8):
  - Department of Internal Medicine, Dr. Kariadi General Hospital, Semarang, Central Java
  - Department of Internal Medicine, Universitas Sebelas Maret (UNS) Hospital, Sukoharjo, Central Java
  - Department of Internal Medicine, Dr. Moewardi Hospital, Surakarta, Central Java
  - Department of Internal Medicine, Budhi Asih Hospital, Jakarta, DKI Jakarta
  - Department of Internal Medicine, Fatmawati General Hospital, Jakarta, DKI Jakarta
  - Department of Internal Medicine, Pasar Rebo Hospital, Jakarta, DKI Jakarta
  - Department of Internal Medicine, Dr. Soetomo General Hospital, Surabaya, Indonesia, Surabaya, East Java
  - Division of Gastroenterology Department of Internal Medicine Faculty of Medicine, University of Indonesia Dr. Cipto Mangunkusumo National General Hospital, Jakarta, Jakarta Special Capital Region

IPD SHARING:
Plan to Share IPD: No